CLINICAL TRIAL: NCT05810584
Title: A Retrospective and Prospective Clinical Study Evaluating Safety and Performance of Revision LR Stem in Total Hip Arthroplasty (THA)
Brief Title: Revision LR Femoral Stem for Hip Replacement
Status: Completed | Type: Observational
Sponsor: Limacorporate S.p.a (Industry)
Responsible Party: Sponsor
Other Study IDs: H-32
Record Dates: First submitted 2023-03-31; First posted 2023-04-12 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Hip Arthropathy; Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Revision LR femoral stem — Revision LR is a modular femoral stem used for hip replacement

SUMMARY:
This is a post-market, monocentric Retrospective and prospective, observational, open-label and baseline clinical study in order to evaluate the performance and safety of Revision LR femoral stem

ELIGIBILITY:
Inclusion Criteria:

* Males and females of any race
* Age ≥ 18 years old
* A diagnosis or condition in the target hip of one or more of the following: Primary tumors or metastasis and relative outcomes; Advanced articular destruction generated by primary degenerative or post-traumatic arthrosis or rheumatoid arthritis;Fracture or avascular necrosis; Congenital or acquired deformity; Failures of previous operations, like osteosynthesis, articular reconstruction, arthrodesis, hemi-arthroplasty or total arthroplasty; Epiphyseal region general trauma, Willingness to comply with prescribed rehabilitation and study evaluation and ability to return for follow-up visits
* Signed study-specific Informed Consent Form

Exclusion Criteria:

* Acute or chronic infections, local or systemic infections,
* Septicaemia
* Persistent acute or chronic osteomyelitis
* Serious muscular, neurological or vascular diseases affecting the concerned limb
* Mass higher than 60 kg

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent a hip arthroplasty with Revision LR stem at Spedali Civili (Brescia) from 1st January 2012 will be screened for the retrospective part of the study. Patients who require a hip arthroplasty with a large femur resection will be screened for the prospective part of the study.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
Revision rate of the femoral component | from baseline to FU 10 Years
  Revision rate of the femoral component for aseptic loosening, not resultant from a tumor recurrence.

SECONDARY OUTCOMES:
Implant stability | from baseline to FU 10 Years
  Implant stability via radiographic assessment of the X-rays at followup, using immediate postoperative X-rays as baseline;
Functionality evaluation | from baseline to FU 10 Years
  Functionality of the patients measured via Harris Hip Score up to last available FU
Incidence of device-related adverse events or serious adverse events. | from baseline to FU 10 Years
  Incidence of device-related adverse events or serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- A.S.S.T Spedali Civili di Brescia, Brescia, Italy